CLINICAL TRIAL: NCT05808257
Title: Superpulsed Thulium Fiber Laser VS. Pulse Modulated High Power Holmium:YAG Laser For Retrograde Intrarenal Surgery
Brief Title: Thulium vs. Hol:YAG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mantu Gupta, Professor of Urology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-22-01521
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Thulium Fibre Laser (TFL) (Experimental): Patients who are randomized to undergo ureteroscopic laser lithotripsy with the Thulium fibre laser (TFL)
  Interventions: Device: Thulium Fibre Laser
- Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) (Experimental): Patients who are randomized to undergo ureteroscopic laser lithotripsy with the Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) laser
  Interventions: Device: Holmium:Yttrium-Aluminum-Garnet

INTERVENTIONS:
Device: Thulium Fibre Laser — The TFL is a relatively new laser in the field of urology. First introduced on the market in 2017, it offers theoretically superior stone dusting qualities and smaller fiber sizes to allow for better irrigation.
  Other Names: TFL
  Arms: Thulium Fibre Laser (TFL)
Device: Holmium:Yttrium-Aluminum-Garnet — The Ho:YAG is currently the most commonly used laser in the field of urology and for the better part of the last 3 decades has been considered the gold standard for laser lithotripsy.
  Other Names: Ho:YAG
  Arms: Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)

SUMMARY:
This is a randomized prospective study to compare stone free rates and operative efficiency of two laser systems used during retrograde intrarenal surgery for kidney stone disease:

1. A superpulsed thulium fiber laser (thulium)
2. A pulse modulated high power holmium laser (Holmium)

DETAILED DESCRIPTION:
This is a randomized prospective study. The purpose is to compare the stone free rate and operative efficiency of two leading contemporary laser systems used during retrograde intrarenal surgery for kidney stone disease. The researchers will compare the following two systems:

1. A superpulsed thulium fiber laser (thulium)
2. A pulse modulated high power holmium laser (Holmium)

The researchers will recruit 82 subjects undergoing single stage unilateral ureteroscopy for renal stones with a volume between >5mm to < 20 mm. Subjects will be randomized to undergo lithotripsy with either Ho:YAG or Thulium lasers.

All subjects will undergo surgical interventions that abide by broadly accepted guidelines and standards of care.

The primary outcome is stone free rate evaluated by postoperative CT scans done 6-12 weeks after surgery.

ELIGIBILITY:
Inclusion criteria:

* Undergoing single stage unilateral RIRS for total stone burden volume >5mm to < 20 mm
* Preoperative CT scan for baseline measurements

Exclusion criteria:

* Anatomic variations: horseshoe kidney, pelvic kidney, ptotic kidney, urinary diversion or ureteral stricture
* Ureteral stent
* Uric acid component >50% on stone analysis
* Prior ureteroscopy within 6 weeks of current surgery
* Irreversible coagulopathy
* Urothelial tumor(s), direct extraction of the stone(s) without needing laser lithotripsy, and failure to reach the stone in the upper urinary tract with the ureteroscope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mantu Gupta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Aggregate results will be published by the investigators in academic journals.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Started | 41 | 41
Completed | 33 | 33
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG) | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.0 [52.3 to 69.8] | 60.0 [45.5 to 72.0] | 60.5 [48.0 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 23 | 25 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 19 | 27 | 46
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 6 | 16
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 27.2 [24.8 to 31.5] | 26.6 [23.4 to 28.6] | 26.8 [24.7 to 29.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stone Free Status
Description: Stone free status as determined by 6-12 week postoperative CT scan to assess laser efficacy
Time Frame: 6-12 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 33 | 33
Participants | 27 | 26

2. Secondary Outcome: Fragmentation Speed
Description: Fragmentation speed is calculated by dividing stone volume by lasing time (mm3/sec). This is a measure of how quickly the laser breaks down the kidney stones.
Time Frame: Intraoperatively (Day 1)
Measure: Median (Inter-Quartile Range); unit: mm3/sec
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 33 | 33
mm3/sec | 0.25 [0.17 to 0.46] | 0.29 [0.18 to 0.39]

3. Secondary Outcome: Lasing Activity
Description: Lasing activity is calculated by dividing lasing time by lithotripsy operative time (%). This measures the percentage of time during surgery that the surgeon is actively using the laser to break down kidney stones.
Time Frame: Intraoperatively (Day 1)
Measure: Median (Inter-Quartile Range); unit: percent of time using laser
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 33 | 33
percent of time using laser | 58.0 [39.6 to 67.3] | 46.1 [36.3 to 55.5]

4. Secondary Outcome: Energy Utilization
Description: Energy utilization is calculated by dividing laser energy by stone volume (J/mm3). This is a measure of how much laser energy is needed to break down a stone.
Time Frame: Intraoperatively (Day 1)
Measure: Median (Inter-Quartile Range); unit: J/mm3
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
Number analyzed (Participants) | 33 | 33
J/mm3 | 13.6 [6.4 to 22.3] | 17.7 [10.2 to 38.7]

ADVERSE EVENTS:
Time Frame: up to 12 weeks postoperative
Arm/Group | Thulium Fibre Laser (TFL) | Holmium:Yttrium-Aluminum-Garnet (Ho:YAG)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT05808257/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05808257/ICF_001.pdf